CLINICAL TRIAL: NCT06430372
Title: Study of Vascular Endothelial Growth Factor A Targeting NIR-II Fluorescence in the Endoscopy of Gastrointestinal Tract
Brief Title: Study of VEGF-A Targeting NIR-II Fluorescence Endoscopy in the Gastrointestinal Tract
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Automation, Chinese Academy of Sciences (Other)
Responsible Party: Principal Investigator, Zhenhua Hu, Professor, Institute of Automation, Chinese Academy of Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: NIR-II-ENDO
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Gastrointestinal Carcinoma; Dysplasia; Gastrointestinal Polyp

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bev-ICG NIR-II Endoscopy (Experimental): The patients will receive a topical administration of probe (Bev-ICG) during the endoscopy. Then fluorescence imaging will be performed to guide the detection.
  Interventions: Drug: Bev-ICG; Device: NIR-II fluorescence endoscopy platform

INTERVENTIONS:
Drug: Bev-ICG — Probe targeting VEGF-A that is topically administrated during the endoscopy
Device: NIR-II fluorescence endoscopy platform — An endoscopic detection device which can detect and visualize NIR-II fluorescent signal during the endoscopy

SUMMARY:
In this study, the investigators are studying new ways to look for abnormal tissues of the gastrointestinal tract during an endoscopy. We are using a VEGF-A targeting fluorescent probe and a NIR-II fluorescent endoscope to help detect abnormal tissues that are hard to see by the naked eye.

The main purposes of this study include:

1. To translate the NIR-II approach into the endoscopy, and understand its advantages and limitations on detecting abnormal tissues in gastrointestinal.
2. To validate whether topical administration of a targeting probe can stick to abnormal tissues and be detected by the NIR-II endoscope.
3. To validate the safety and effectiveness of the topical administration of VEGF-A targeting probes for clinical application.

ELIGIBILITY:
Inclusion Criteria:

* Known or suspected gastrointestinal lesions.
* Scheduled for a clinically-indicated endoscopy.
* Mentally competent person, 18 years or older.
* Approved to sign the informed consent.
* Adequate potential for follow-up.

Exclusion Criteria:

* Subjects with known allergy or negative reaction to ICG or derivatives.
* Undesirable function of heart, lung, kidney, or any other organs.
* Enrolled in other trials in the past 3 months.
* Pregnant or trying to conceive.
* Unable to tolerate an endoscopy.
* Medical or psychiatric conditions that compromise the patient's ability to give informed consent.
* The researchers considered inappropriate to be included.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Validation of NIR-II endoscope and probe targeting VEGF-A | During endoscopy
  Demonstrate the feasibility of using the NIR-II endoscope and VEGF-A targeting fluorescent probe to image abnormal tissues of the gastrointestinal tract.

CONTACTS AND LOCATIONS:
Locations (1):
- Lidan Fu, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No